CLINICAL TRIAL: NCT06054373
Title: The Distribution of Immunoglobulin Isotype in Polyclonal Hypergammaglobulinemia in Systemic and Autoimmune Diseases
Acronym: ISOHYPE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Binding site (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0116
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Polyclonal Hypergammaglobulinemia; Autoimmune Diseases
Keywords: Polyclonal Hypergammaglobulinemia; Autoimmune Diseases; immunoglobulin isotypes
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Polyclonal hypergammaglobulinaemia is characterized by increased levels of immunoglobulins and is a common feature observed in various diseases such as autoimmune diseases, chronic infectious diseases or lymphoid hemopathy. Some autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis or Sjögren's syndrome are frequently associated with polyclonal hypergammaglobulinaemia. Recent data have suggested that the distribution of immunoglobulin isotypes in polyclonal hypergammaglobulinaemia may be disease-specific. However, isotype repartition in polyclonal hypergammaglobulinaemia remains poorly understood.

The investigators will investigate the distribution of immunoglobulin isotype in patients with autoimmune disease and polyclonal hypergammaglobulinaemia. Moreover, the investigators will evaluate the isotype repartition as predictor of lymphoma or monoclonal gammopathy among patients with autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > 18 years old
* patients with one of the following diseases: systemic lupus erythematosus, rheumatoid arthritis, Sjögren's syndrome, autoimmune hepatitis, sarcoidosis or lymphoma.

Exclusion Criteria:

* Age < 18 years;
* chronic viral hepatitis;
* HIV infection, syphilis,
* tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diagnosis of various autoimmune diseases and polyclonal hypergammaglobulinaemia. Medical records from 2004 to 2018 were reviewed to identify eligible patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
distribution of immunoglobulin isotypes | one day
  distribution of immunoglobulin isotypes in polyclonal hypergammaglobulinaemia associated with autoimmune and systemic diseases (systemic lupus erythematosus, rheumatoid arthritis, Gougerot-Sjögren syndrome, sarcoidosis)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No